CLINICAL TRIAL: NCT07360548
Title: 18F-fluoro-ethyl-tyrosine (18FET) PET for Difficult Clinical Situations in Functional Pituitary Adenoma. A Prospective, Single Arm, Single Center Study
Brief Title: Study of 18FET PET in Functional Pituitary Adenomas With Indeterminate MRI Findings
Acronym: FET-PIT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025_0205
Record Dates: First submitted 2025-12-10; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Functional Pituitary Adenomas
Keywords: PET-18 Fluoro ethyl tyrosine; Functional pituitary adenoma; Indeterminate MRI
MeSH Terms: interventions — (18F)fluoroethyltyrosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): The investigative procedure used is 18FET PET, which will be the only difference from the usual care.
  The study data (clinical observations, laboratory results, imaging results) will be collected by the various study investigators during a consultation and/or via the Lille University Hospital computer server.
  Performance of the 18FET PET scan in the Nuclear Medicine Department. The experimental drug is [18F]Fluoroethyl-L-tyrosine, produced in accordance with Good Manufacturing Practices (GMP) guidelines and marketed under the name IASOglio by Curium PET France. The maximum activity for an adult is to 250 MBq. This activity must be administered by direct intravenous injection.
  Shelf life: 14 hours from the end of synthesis. After first use or after dilution, the product can be stored for up to 8 hours without exceeding the expiry date of 14 hours from the end of synthesis.
  Interventions: Drug: fluoroethyl-L tyrosine (18F)

INTERVENTIONS:
Drug: fluoroethyl-L tyrosine (18F) — The protocol consists of a single arm involving the administration of the radiopharmaceutical 18FET (IASOglio).
  This will be administered once during the study, directly intravenously with an activity of 200 +/- 15MBq, as recommended by the European EANM/EANO/RANO guidelines and used in retrospective studies investigating the contribution of 18FET in AP. Included patients will have fasted for at least 4 hours beforehand. PET image acquisition will begin as soon as the radiopharmaceutical is injected.
  Other Names: IASOglio 2 GBq/mL : Marketing authorization number : 34009 550 105 1 7 (15mL) / 34009 550 105 2 4 (25 mL)

SUMMARY:
Pituitary adenomas (PAs) are common benign tumors, but their potential for tumor aggression and hormone secretion make them serious tumors. In particular, patients with secreting tumors [prolactinomas (prolactin secretion), acromegaly (growth hormone), Cushing's disease (ACTH), thyrotropic adenomas (TSH)] have increased morbidity and mortality. They may be small and/or undetectable by magnetic resonance imaging (MRI), the current gold standard for morphological evaluation of pituitary lesions. The diagnosis of recurrence in a patient who has already undergone surgery also raises the problem of distinguishing between a lesion and postoperative remodeling. The detection of these tumors therefore represents a significant challenge in guiding therapeutic management.Nuclear medicine could solve this challenge, particularly radiopharmaceuticals (MRPs) used in PET (positron emission tomography) combined with CT scans. A few studies have evaluated MRPs in the context of APs, with those targeting amino acid metabolism proving to be the most promising, particularly carbon-11-labeled methionine (11C-MET). In retrospective studies only, 11C-MET PET has shown excellent performance in all situations where MRI fails (detection rate >80%), but the extremely short half-life of 11C requires heavy infrastructure, limiting its access in routine clinical practice.18Fluoroethyl-Tyrosine (18FET) is also a PET MRP targeting amino acid metabolism used in France in neuro-oncology with performance equivalent to 11C-MET, and which has the advantage of being available daily in all nuclear medicine centers.

The performance of 18FET in APs is almost unknown, with only two retrospective studies recently published, including 22 patients with Cushing's disease on the one hand and 17 patients with prolactinoma on the other: The detection rates were particularly interesting (82% and 100% respectively), but it is imperative to confirm these data prospectively and to evaluate the performance of this MRP in other functional types, which is therefore the purpose of this study.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female
* Aged 18 years or older
* Suspected of having a functional pituitary adenoma (prolactinoma - Cushing's disease - acromegaly - thyrotropic adenoma), de novo or recurrence/persistence
* With indeterminate pituitary MRI
* Patient covered by social security
* Patient willing to comply with all study procedures and duration
* Patient eligible for surgery and/or radiotherapy in case of positive 18FET PET scan

Exclusion Criteria:

* Pregnancy
* Known hypersensitivity to radiopharmaceuticals
* Administrative reasons: inability to receive informed information, inability to participate in the entire study, lack of coverage by the social security system, refusal to sign the consent form
* Contraindication to surgery and radiotherapy in the case of positive 18FET PET
* Patients who are active alcohol users
* Patients suffering from liver disease or severe uncontrolled epilepsy
* Patients deprived of their liberty (guardianship, curatorship, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Describe the ability of 18FET PET to detect functional pituitary adenomas in patients with de novo, recurrent, or persistent functional AP when pituitary MRI is non-contributive. | 2 months +/- 2 months
  Frequency of patients for whom PET would be useful among patients with a positive 18FET PET result.The gold standard will be defined by the pathological examination of the surgical specimen in the case of surgery, or by the possibility of stopping or gradually reducing medical treatment while maintaining normalized hormone secretion in the case of radiotherapy.

SECONDARY OUTCOMES:
Describe the frequency of patients positive for 18FET PET in patients with de novo, recurrent, or persistent functional AP when pituitary MRI is non-contributive. | 2 months +/- 2 months
  Frequency of patients with positive 18FET PET scans.
Describe SUVmax based on the 18FET PET scan result | 2 months +/- 2 months
  SUVmax (g/mL) based on the result of the 18FET PET scan (patients negative on the 18FET PET scan, patients positive on the 18FET PET scan and successfully treated, and patients positive on the 18FET PET scan but not treated or treatment failure).
Describe Adenoma/healthy brain ratio based on the 18FET PET scan result | 2 months +/- 2 months
  Based on the result of the 18FET PET scan (patients negative on the 18FET PET scan, patients positive on the 18FET PET scan and successfully treated, and patients positive on the 18FET PET scan but not treated or treatment failure).
Describe kinetic parameters based on the 18FET PET scan result. | 2 months +/- 2 months
  Kinetic parameters (time to peak in minutes) based on the result of the 18FET PET scan (patients negative on the 18FET PET scan, patients positive on the 18FET PET scan and successfully treated, and patients positive on the 18FET PET scan but not treated or treatment failure).
Measure the concordance of the 18FET PET scan results between three readers. | 2 months +/- 2 months
  Concordance will be measured by the Krippendorf coefficient.
Describe the proportion of patients who, following 18FET PET, received therapeutic treatment targeting the adenoma (surgery and/or external radiation therapy). | 1 year +/- 2 months
  Frequency of patients undergoing surgery and frequency of patients undergoing radiation therapy among patients who tested positive on 18FET PET scans.

IPD SHARING:
Plan to Share IPD: No